CLINICAL TRIAL: NCT00278421
Title: Randomized Study Comparing 4 and 6 Cycles of Chemotherapy With CHOP (Cyclophosphamide, Doxorubicin, Vincristine and Prednisone) at 21-day Intervals, Both With 6 Cycles of Immunotherapy With the Monoclonal Anti-CD20-Positive B-Cell Lymphoma Aged 18-60 Years Having no Risk Factor (Age-Adjusted IPI=0) and No Large Tumor Mass (Diameter <7,5cm) [FLYER 6-6-6-4 Study]
Brief Title: Rituximab and Combination Chemotherapy in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German High-Grade Non-Hodgkin's Lymphoma Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000459685; DSHNHL-2004-2; EU-205110; EUDRACT-2005-00521738; DSHNHL-FLYER-6664
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage I grade 3 follicular lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; nodal marginal zone B-cell lymphoma; anaplastic large cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II mantle cell lymphoma; stage I adult Burkitt lymphoma; stage I mantle cell lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional: 6 R-CHOP-21 (Active Comparator): Arm I: Patients receive R-CHOP immunochemotherapy comprising rituximab IV, cyclophosphamide IV over 15 minutes, doxorubicin hydrochloride IV, and vincristine IV on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo restaging of their disease. Patients with disease progression proceed to salvage therapy off study. All other patients receive 3 more courses of R-CHOP.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate
- Interventional: 4 R-CHOP-21 + 2 x R (Active Comparator): Arm II: Patients receive R-CHOP as in arm I. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo restaging of their disease. Patients with disease progression proceed to salvage therapy off study. All other patients receive 1 more course of R-CHOP followed by 2 courses of rituximab alone.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving rituximab together with combination chemotherapy may kill more cancer cells. It is not yet known which schedule of rituximab and combination chemotherapy is more effective in treating non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying two different schedules of rituximab and combination chemotherapy to compare how well they work in treating patients with aggressive B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of 2 different schedules of immunochemotherapy comprising rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone in patients with previously untreated, low-risk, aggressive B-cell non-Hodgkin's lymphoma.
* Compare acute and chronic side effects in patients treated with these regimens.
* Compare time to treatment failure in patients treated with these regimens.

Secondary

* Compare the time to progression in patients treated with these regimens.
* Compare the overall and disease-free/relapse-free survival of patients treated with these regimens.
* Compare the complete response rate in patients treated with these regimens.
* Compare the tumor control in patients treated with these regimens.
* Compare the safety of these regimens in these patients.
* Compare the pharmacoeconomics of these regimens.
* Compare patient adherence to these regimens.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

All patients are given the option of receiving a 1-week course of pretreatment therapy comprising vincristine IV once on day -6 and oral prednisone once daily on days -6 to 0.

* Arm I: Patients receive R-CHOP immunochemotherapy comprising rituximab IV, cyclophosphamide IV over 15 minutes, doxorubicin hydrochloride IV, and vincristine IV on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo restaging of their disease. Patients with disease progression proceed to salvage therapy off study. All other patients receive 3 more courses of R-CHOP.
* Arm II: Patients receive R-CHOP as in arm I. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo restaging of their disease. Patients with disease progression proceed to salvage therapy off study. All other patients receive 1 more course of R-CHOP followed by 2 courses of rituximab alone.

All patients undergo final restaging after 6 courses of rituximab. Patients with disease progression, stable disease, or partial response proceed to salvage therapy off study.

After completion of study treatment, patients are followed periodically for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 622 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive B-cell non-Hodgkin's lymphoma, including the following subtypes:

  * Grade 3 follicular lymphoma
  * Diffuse B-cell lymphoma, including diffuse large cell lymphoma with any of the following variants:

    * Centroblastic
    * Immunoblastic
    * Plasmablastic
    * Anaplastic large cell
    * T-cell-rich B-cell lymphoma
  * Primary effusion lymphoma
  * Intravascular B-cell lymphoma
  * Primary mediastinal B-cell lymphoma
  * Burkitt's or Burkitt-like lymphoma
  * Mantle cell lymphoma (blastoid)
  * Aggressive marginal zone lymphoma (monocytoid)
* Previously untreated disease
* CD20-positive disease
* International Prognostic Index (IPI) score 0
* No bulky disease

  * Largest single or conglomerate tumor < 7.5 cm in diameter
* No mucosa-associated lymphoid tissue (MALT) lymphoma
* No CNS involvement of lymphoma (intracerebral, meningeal, or intraspinal)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 2,500/mm^3
* Lactate dehydrogenase normal
* Not pregnant or lactating
* Fertile patients must use effective contraception during and for 1 year after study participation
* Negative pregnancy test
* No known hypersensitivity to the study medications
* No known HIV-positivity
* No active hepatitis infection
* No impaired left ventricular function
* No severe cardiac arrhythmias
* No other impaired organ function
* No other serious disorder
* No other malignancy within the past 5 years except carcinoma in situ or basal cell skin cancer

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy
* No prior immunosuppressive treatment with cytostatics
* No planned radiotherapy to extranodal involvement
* No concurrent participation in other treatment studies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 592 (Actual)
Dates: Start 2005-11; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) measured from day 1 of course 1 of Cyclophosphamide, Doxorubicin, Vincristine and Prednisone (CHOP) therapy up to 3 years on study with life-long follow-up | through study completion

SECONDARY OUTCOMES:
Complete response (CR) rate duration until first relapse | through study completion
Progression rate during treatment | through study completion
Survival | through study completion
Tumor control measured from day 1 of course 1 of CHOP therapy (non-tumor related events are censored) | through study completion
Disease-free survival measured from day 1 of course 1 of CHOP therapy | through study completion
Safety (adverse events, serious adverse events) assessed at 3 months after treatment | through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Michael G.M. Pfreundschuh, MD †, Study Chair — Universitaetsklinikum des Saarlandes; Viola Poeschel, MD, Study Director — Study Office Homburg
Locations (78):
- Germany (74):
  - Haematologisch Onkologische Praxis, Aachen
  - Klinikum Augsburg, Augsburg
  - Klinikum Bayreuth, Bayreuth
  - Haematologisch-Onkologische Schwerpunktpraxis - Weilheim, Berlin
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Franziskus Hospital, Bielefeld
  - Augusta-Kranken-Anstalt gGmbH, Bochum
  - Staedtisches Klinikum Braunschweig, Braunschweig
  - DIAKO Ev. Diakonie Krankenhaus gGmbH, Bremen
  - Hospital Kuchwald Chemnitz, Chemnitz
  - Praxis Fuer Haematologie Internistische Onkologie, Cologne
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Carl - Thiem - Klinkum Cottbus, Cottbus
  - Praxis Dr. Rheinhold Siegmund - Dr. Matthias Penke, Damme
  - Klinikum Dortmund, Dortmund
  - Hans - Susemihl - Krankenhaus, Emden
  - St. Antonius Hospital, Eschweiler
  - Universitaetsklinikum Essen, Essen
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum Fulda, Fulda
  - Saint Josef Hospital, Gelsenkirchen
  - Universitaetsklinikum Goettingen, Göttingen
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Kreiskrankenhaus Gummersbach GMBH, Gummersbach
  - St. Marien Hospital - Katholisches Krankenhaus Hagen gGmbH, Hagen
  - St. Sixtus Hospital, Haltern
  - Asklepios Klinik St. Georg, Hamburg
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Haematologisch-Onkologische Praxis Altona, Hamburg
  - St. Marien-Hospital Hamm - Klinik Knappenstrasse, Hamm
  - Evangelische Krankenhaus Hamm, Hamm
  - Medizinische Hochschule Hannover, Hanover
  - Ruprecht - Karls - Universitaet Heidelberg, Heidelberg
  - St. Bernward Krankenhaus, Hildesheim
  - Universitaetsklinikum des Saarlandes, Homburg
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - St. Vincentius - Kliniken, Karlsruhe
  - Klinikum Kempten Oberallgaeu, Kempten
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Caritas - Krakenhaus Lebach, Lebach
  - Klinikum Lippe - Lemgo, Lemgo
  - St. Vincenz Hospital Limburg, Limburg
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen am Rhein
  - Kreiskrankenhaus Luedenscheid, Lüdenscheid
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - III Medizinische Klinik Mannheim, Mannheim
  - Universitaetsklinikum Giessen und Marburg GmbH - Marburg, Marburg
  - Krankenhaus Ludmillenstift, Meppen
  - Krankenhaus Maria Hilf GmbH, Mönchengladbach
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Klinikum Schwaebisch Gmuend Stauferklinik, Mutlangen
  - Haematologisch - Onkologische Gemeinschaftspraxis - Muenster, Münster
  - Medizinische Klinik und Poliklinik A - Universitaetsklinikum Muenster, Münster
  - Onkologische Schwerwpunktpraxis Dr. Ladda, Neumarkt
  - Lukaskrankenhaus Neuss, Neuss
  - Schlossbergkliniken Oberstaufen, Oberstaufen
  - Klinikum Oldenburg, Oldenburg
  - Pforzheim
  - Klinikum Ernst Von Bergmann, Potsdam
  - Prosper-Hospital Recklinghausen, Recklinghausen
  - Rostock
  - St. Marien - Krankenhaus Siegen GMBH, Siegen
  - Diakonie Klinikum Stuttgart, Stuttgart
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
  - Universitaetsklinikum Tuebingen, Tübingen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - St. Marienhospital - Vechta, Vechta
  - Onkologische Schwerpunktpraxis, Wendlingen
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Helios Kliniken Wuppertal University Hospital, Wuppertal
- Rabin Medical Center - Beilinson Campus, Petah Tikva, Israel
- Italy (3):
  - Ospedale Civile - Piacenza, Piacenza
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Cellulari ed Ematologia Sapienza, Roma

REFERENCES:
- [Derived] Poeschel V, Held G, Ziepert M, Witzens-Harig M, Holte H, Thurner L, Borchmann P, Viardot A, Soekler M, Keller U, Schmidt C, Truemper L, Mahlberg R, Marks R, Hoeffkes HG, Metzner B, Dierlamm J, Frickhofen N, Haenel M, Neubauer A, Kneba M, Merli F, Tucci A, de Nully Brown P, Federico M, Lengfelder E, di Rocco A, Trappe R, Rosenwald A, Berdel C, Maisenhoelder M, Shpilberg O, Amam J, Christofyllakis K, Hartmann F, Murawski N, Stilgenbauer S, Nickelsen M, Wulf G, Glass B, Schmitz N, Altmann B, Loeffler M, Pfreundschuh M; FLYER Trial Investigators; German Lymphoma Alliance. Four versus six cycles of CHOP chemotherapy in combination with six applications of rituximab in patients with aggressive B-cell lymphoma with favourable prognosis (FLYER): a randomised, phase 3, non-inferiority trial. Lancet. 2019 Dec 21;394(10216):2271-2281. doi: 10.1016/S0140-6736(19)33008-9. PMID 31868632